CLINICAL TRIAL: NCT02372578
Title: A Phase 2a Randomized, Double-Blind, Multicenter, Placebo and Active Controlled Study to Assess Analgesic Efficacy and Safety of ASP3662 in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: Study to Assess Analgesic Efficacy and Safety of ASP3662 in Subjects With Painful Diabetic Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to futility analysis.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3662-CL-0049
Record Dates: First submitted 2015-02-21; First posted 2015-02-26 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Painful Diabetic Peripheral Neuropathy (PDPN)
Keywords: Painful diabetic peripheral neuropathy (PDPN); ASP3662
MeSH Terms: interventions — ASP3662; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ASP3662 (Experimental): ASP3662 once daily (QD) and pregabalin placebo 3 times daily (TID) for Weeks 1 - 6. ASP3662 placebo QD and pregabalin placebo TID for Week 7.
  Interventions: Drug: ASP3662; Drug: ASP3662 placebo; Drug: pregabalin placebo
- pregabalin (Active Comparator): pregabalin TID and ASP3662 placebo QD for Weeks 1 - 7.
  Interventions: Drug: pregabalin; Drug: ASP3662 placebo
- Placebo (Placebo Comparator): ASP3662 placebo QD and pregabalin placebo TID for Weeks 1 - 7.
  Interventions: Drug: ASP3662 placebo; Drug: pregabalin placebo

INTERVENTIONS:
Drug: ASP3662 — oral
  Arms: ASP3662
Drug: pregabalin — oral
  Arms: pregabalin
Drug: ASP3662 placebo — oral
Drug: pregabalin placebo — oral
  Arms: ASP3662; Placebo

SUMMARY:
The purpose of this study is to assess analgesic efficacy of ASP3662 relative to placebo in subjects with painful diabetic peripheral neuropathy (PDPN) as well as assess the safety and tolerability of ASP3662 relative to placebo.

The analgesic effect is evaluated by measuring percent responders, change in daily worst pain score, change in average daily pain score, Patient Global Impression of Change (PGIC) and Clinical Global Impression of Change (CGIC).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a BMI ≤ 40.
* Subject has all of the following:

  1. Established diagnosis of diabetes (Type I or II) with painful diabetic peripheral neuropathy and glycosylated hemoglobin (HgbA1c) ≤ 9.5% at Screening or Randomization.
  2. Stable diabetic drug regimen for at least 3 months prior to Screening.
  3. At least a 1 year history of PDPN.
  4. Diagnosis of PDPN to be confirmed by a score of ≥ 3 on the Michigan Neuropathy Screening Instrument (MNSI) at Screening.
* Subject has pain intensity score(s) ≥ 4 or ≤ 9 on an 11-point numeric pain rating scale (NPRS) at Screening Visit and prior to Randomization.
* Subject agrees to complete pain diaries and is complaint with the daily pain recording prior to Randomization as defined by the completion of a minimum of 5 of 7 daily pain ratings, 3 of which are required in the last 4 days.
* Subject's anti-diabetic regimen is anticipated to be stable throughout the study.
* Subject must be willing to washout of all medications currently being taken for his/her PDPN (chronic and occasional/as needed) and remain off of those pain medications while participating in the study.

Exclusion Criteria:

* Subject has received prior treatment with pregabalin for PDPN and was considered unresponsive or intolerant.
* Subject has tried and failed 3 or more drugs to treat PDPN within the past 3 years. Drugs must have been administered at therapeutic doses and have been administered for an adequate period of time.
* Subject has a known hypersensitivity to ASP3662, pregabalin, gabapentin or acetaminophen, or their formulation components.
* Subject has significant pain (moderate or above) due to causes other than PDPN.
* Subject has a history of painful peripheral neuropathy due to a cause other than diabetes.
* Subject has any lower extremity amputation
* Subject has a current or previous foot ulcer within the past 3 months as described by medical history and/or medical examination.
* Subject has an active malignancy or a history of malignancy (except for treated non-melanoma skin cancer) within 5 years.
* Subject has clinically significant abnormalities in clinical chemistry, hematology, or urinalysis, or a serum creatinine at Screening.
* Subject has creatinine clearance < 60 mL/min (estimated from serum creatinine, body weight, age, and sex using the Cockcroft and Gault equation) at Screening.
* Subject tests positive for hepatitis B surface antigen (HBsAg) or hepatitis C antibody at Screening or has a known history of a positive test for human immunodeficiency virus (HIV) infection.
* Subject has a positive drug screen for alcohol or drugs of abuse at Screening and/or Randomization. Subjects who are on low doses of benzodiazepines for sleep with a legitimate prescription will be allowed into the study. In addition, subjects with a positive drug screen at Randomization will be excluded.
* Subject is currently using protocol specified non-permitted medications including OTC products and is unable or does not choose to discontinue them.
* Subject has planned an elective surgery during planned study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in mean 24-hour average pain intensity as reported on the NPRS | Baseline to Week 6/ End of Treatment (EOT)
  Numerical Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Percentage of Responders in mean 24-hour average pain intensity score | Baseline to Week 6/ EOT
Change from Baseline in mean of 24-hour average pain intensity score | Baseline to Weeks 1, 2, 3, 4, 5 and 6
Change from Baseline in mean daily worst pain score | Baseline to Week 6/ EOT
Change from Baseline in mean daily average pain score | Baseline to Week 6/ EOT
Patient Global Impression Change (PGIC) | Week 6/ EOT
Clinical Global Impression of Change (CGIC) | Week 6/ EOT

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (37):
- United States (37):
  - Site US10001, Anniston, Alabama
  - Site US10039, Phoenix, Arizona
  - Site US10054, Fresno, California
  - Site US10020, Lomita, California
  - Site US10047, Santa Monica, California
  - Site US10017, Tustin, California
  - Site US10055, Walnut Creek, California
  - Site US10053, Fairfield, Connecticut
  - Site US10005, Boynton Beach, Florida
  - Site US10023, Bradenton, Florida
  - Site US10018, Clearwater, Florida
  - Site US10019, DeLand, Florida
  - Site US10004, Homestead, Florida
  - Site US10042, Jacksonville, Florida
  - Site US10007, Jupiter, Florida
  - Site US10041, Miami Lakes, Florida
  - Site US10046, Orlando, Florida
  - Site US10008, Ormond Beach, Florida
  - Site US10003, Oviedo, Florida
  - Site US10049, The Villages, Florida
  - Site US10009, Aurora, Illinois
  - Site US10036, Chicago, Illinois
  - Site US10025, Evansville, Indiana
  - Site US10064, Metairie, Louisiana
  - Site US10051, Boston, Massachusetts
  - Site US10026, New Bedford, Massachusetts
  - Site US10063, Quincy, Massachusetts
  - Site US10043, Hazelwood, Missouri
  - Site US10013, Kettering, Ohio
  - Site US10014, Duncansville, Pennsylvania
  - Site US10015, Greer, South Carolina
  - Site US10034, Austin, Texas
  - Site US10040, Houston, Texas
  - Site US10032, San Antonio, Texas
  - Site US10031, San Antonio, Texas
  - Site US10033, Salt Lake City, Utah
  - Site US10045, Renton, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Studies conducted with product indications or formulations that remain in development are assessed after study completion to determine if Individual Participant Data can be shared. The plan to share Individual Participant Data is based on the status of product approval or termination of the compound, in addition to other study-specific criteria described on www.clinicalstudydatarequest.com under "Sponsor Specific Details for Astellas."

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=297